CLINICAL TRIAL: NCT06081465
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Orally Administered VG290131 in Healthy Adult Subjects
Brief Title: A Phase I Study of Single and Multiple Doses of VG290131 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Vimgreen Pharmaceuticals, Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: VG290131-AU-001
Record Dates: First submitted 2023-09-30; First posted 2023-10-13 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: The study consists of three parts: a single ascending dose (SAD) part, a multiple ascending dose (MAD) part and a food effect (FE) part. The FE study is incorporated as part of the SAD study. Approximately 86 subjects will be enrolled in the study.
  SAD+FE study: 6 cohorts (1, 5, 25, 50, 100, and 200 mg), 8 subjects in each cohort, except that there are 14 subjects in the 5 mg cohort, which is the FE study cohort.
  MAD study: 4 cohorts (1, 5, 25, and 100 mg), 8 subjects in each cohort.
Who Masked: Participant, Investigator
Masking Description: Eligible subjects will be sequentially enrolled cohort by cohort. In each cohort, subjects will be randomized to receive VG290131 or matching placebo, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- SAD Cohort 1 (Experimental): In SAD Cohort 1, 8 subjects will be randomized to receive a single dose of VG290131 (1 mg) (n=6) or matching placebo (n=2), respectively. To ensure the safety of the subjects, two sentinel subjects will be enrolled first: one subject will be randomized to receive VG290131, and the other subject will be randomized to receive a placebo. After the investigator reviews safety/tolerability information available on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in the cohort will be randomized to receive VG290131 (n=5) and placebo (n=1).
  Interventions: Drug: VG290131
- SAD Cohort 2 (FE Study) (Experimental): SAD Cohort 2 (FE study) is a two-sequence, two-period crossover study. A total of 14 healthy subjects will be randomized to two dosing sequences in a 1:1 ratio. Subjects in sequence 1 will receive a single dose of VG290131 (5 mg) or placebo under fasted condition in Period 1 and under fed condition in Period 2. Subjects in sequence 2 will be administered under fed condition in Period 1 and under fasted condition in Period 2. There will be a 7-day washout between the two dosing periods. Two sentinel subjects will be enrolled in the two dosing sequences of Period 1, respectively: one subject will be randomized to receive VG290131 (5 mg), and the other subject will be randomized to receive placebo. After the investigator reviews safety/tolerability information on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in that sequences will be randomized to receive VG290131 (n=4) and placebo (n=1). No sentinel subjects in Period 2.
  Interventions: Drug: VG290131
- SAD Cohort 3 (Experimental): In SAD Cohort 3, 8 subjects will be randomized to receive a single dose of VG290131 (25 mg) (n=6) or matching placebo (n=2), respectively. To ensure the safety of the subjects, two sentinel subjects will be enrolled first: one subject will be randomized to receive VG290131, and the other subject will be randomized to receive a placebo. After the investigator reviews safety/tolerability information available on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in the cohort will be randomized to receive VG290131 (n=5) and placebo (n=1).
  Interventions: Drug: VG290131
- SAD Cohort 4 (Experimental): In SAD Cohort 4, 8 subjects will be randomized to receive a single dose of VG290131 (50 mg) (n=6) or matching placebo (n=2), respectively. To ensure the safety of the subjects, two sentinel subjects will be enrolled first: one subject will be randomized to receive VG290131, and the other subject will be randomized to receive a placebo. After the investigator reviews safety/tolerability information available on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in the cohort will be randomized to receive VG290131 (n=5) and placebo (n=1).
  Interventions: Drug: VG290131
- SAD Cohort 5 (Experimental): In SAD Cohort 5, 8 subjects will be randomized to receive a single dose of VG290131 (100 mg) (n=6) or matching placebo (n=2), respectively. To ensure the safety of the subjects, two sentinel subjects will be enrolled first: one subject will be randomized to receive VG290131, and the other subject will be randomized to receive a placebo. After the investigator reviews safety/tolerability information available on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in the cohort will be randomized to receive VG290131 (n=5) and placebo (n=1).
  Interventions: Drug: VG290131
- SAD Cohort 6 (Experimental): In SAD Cohort 6, 8 subjects will be randomized to receive a single dose of VG290131 (200 mg) (n=6) or matching placebo (n=2), respectively. To ensure the safety of the subjects, two sentinel subjects will be enrolled first: one subject will be randomized to receive VG290131, and the other subject will be randomized to receive a placebo. After the investigator reviews safety/tolerability information available on the sentinel subjects after 24 h and no significant safety issues are observed, the subsequent subjects in the cohort will be randomized to receive VG290131 (n=5) and placebo (n=1).
  Interventions: Drug: VG290131
- MAD Cohort 1 (Experimental): In MAD Cohort 1, 8 subjects will be randomized 3:1 to receive a once or twice daily dose of VG290131 (1 mg) (n=6) or matching placebo (n=2) for 7 consecutive days depending on the PK profiles of the SAD study, respectively.
  Interventions: Drug: VG290131
- MAD Cohort 2 (Experimental): In MAD Cohort 1, 8 subjects will be randomized 3:1 to receive a once or twice daily dose of VG290131 (5 mg) (n=6) or matching placebo (n=2) for 7 consecutive days depending on the PK profiles of the SAD study, respectively.
  Interventions: Drug: VG290131
- MAD Cohort 3 (Experimental): In MAD Cohort 1, 8 subjects will be randomized 3:1 to receive a once or twice daily dose of VG290131 (25 mg) (n=6) or matching placebo (n=2) for 7 consecutive days depending on the PK profiles of the SAD study, respectively.
  Interventions: Drug: VG290131
- MAD Cohort 4 (Experimental): In MAD Cohort 1, 8 subjects will be randomized 3:1 to receive a once or twice daily dose of VG290131 (100 mg) (n=6) or matching placebo (n=2) for 7 consecutive days depending on the PK profiles of the SAD study, respectively.
  Interventions: Drug: VG290131

INTERVENTIONS:
Drug: VG290131 — The study drug and matching placebo will be administered orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I study to evaluate the safety, tolerability and PK profiles of orally administered VG290131 in healthy subjects. The main questions it aims to answer are:

1. The safety and tolerability of VG290131 when administered orally as a single dose and multiple doses in healthy subjects.
2. The pharmacokinetic (PK) profiles of VG290131 and the food effect on the PK profiles of VG290131 in healthy subjects.

Approximately 86 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria are met:

1. Willing to comply with protocol required visit schedule and visit requirements and provide written ICF;
2. Healthy adult male and female subjects, aged 18 to 45 years of age (inclusive) at the time of signing the ICF;
3. Body mass index between 18.0 and 32.0 kg/m2, inclusive;
4. Considered medically healthy as determined by the investigator, based on medical history and clinical evaluations including physical examination, clinical laboratory tests, vital sign measurements, and 12-Lead ECG;
5. Male subjects must agree to practice true abstinence; be surgically sterilized (performed at least 6 months prior to screening and documented to no longer produce sperm - verbal confirmation through medical history review acceptable); or agree to use a condom plus effective contraception methods for their female partner, if of childbearing potential, from the signing of ICF to 3 months after the last dose of IMPs and refrain from donating sperm during this period. These contraception requirements do not apply if the male subject is in an exclusively same sex relationship;
6. Female subjects are eligible to participate if they are not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

   * Women of non-childbearing potential (WONCBP), defined as surgically sterile (hysterectomy, bilateral salpingectomy, bilateral tubal ligation or bilateral oophorectomy - verbal confirmation through medical history review acceptable) or postmenopausal (no menses for 12 months and confirmed by follicle stimulating hormone [FSH] level ≥40 mlU/mL);
   * WOCBP and agree to practice true abstinence or agrees to use a highly effective method of contraceptions consistently from the signing of ICF to 3 months after the last dose of investigational medicinal products [IMPs] and refrain from donating eggs during this period. And WOCBP must have a negative serum and/or urine pregnancy test result within 7 days prior to the first dose of IMPs.
   * Subject is in an exclusively same-sex relationship.

Exclusion Criteria:

A subject meeting any of the following exclusion criteria will not be allowed to participate in this study:

1. Ascertained or presumptive hypersensitivity (including allergies) to any ingredient of the VG290131; history of other significant allergies or anaphylaxis, as determined by the investigator;
2. Considered by the investigator to be ineligible for the study due to a history of or current condition of significant metabolic or endocrine, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, immunological, neurological, or psychiatric disorders with clinical manifestations;
3. Active or history of serious mental illness or psychiatric disorder, including but not limited to schizophrenia, bipolar disorder, or severe depression, which require current pharmacological intervention;
4. History of stomach or intestinal surgery or resection diseases including but not limited to, gastric band/gastric resection and/or intestinal resection and/or duodenal disease (i.e. celiac disease) which may potentially alter absorption and/or excretion of VG290131 (except for an appendectomy);
5. Used drugs or substances known to be inducers or inhibitors of cytochrome P450 enzymes or P-glycoprotein (P-gp) substrates within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMPs;
6. Used prescription or over-the-counter (OTC) drugs (with the exception of hormonal contraception, menopausal hormone replacement therapy or occasional analgesics such as Paracetamol [1 g per dose and maximum 2-4 g per day], Ibuprofen and standard daily vitamins etc. in short term at the Investigator's discretion), within 14 days or 5 half-lives (whichever is longer) prior to the first dose of IMPs;
7. Participated in any other investigational trials or has been exposed to other investigational drugs within 28 days or 5 half-lives of the previously administered investigational drug, whichever is longer, prior to the first dose of IMPs;
8. Smoking ≥ 5 cigarettes per day (or an equivalent amount of any other nicotine-containing products) within 6 months before screening or unable to stop smoking during the study;
9. Alcohol consumption of > 21 units per week for males and > 14 units per week for females within the 6 months before screening (1 unit=360 mL of beer or 45 mL of spirits with an alcohol content of ≥ 40% or 150 mL of wine) or a positive result of alcohol breath test on admission or unable to abstain from consuming alcohol from 24 h prior to admission, until completion of the end of study (EOS) visit;
10. History of drug abuse within the 12 months before screening or a positive result of drug abuse test at screening;
11. Consumption of any nutrients known to modulate cytochrome P450 enzymes or P-gp substrates activity (eg, grapefruit, pomelo, mango, star fruit, Seville [blood] orange products, caffeine or xanthine-containing food or beverages) within 72 h before the first dose of IMPs;
12. Clinically significant laboratory abnormalities, as determined by the Investigator, including but not limited to (If the results are beyond the normal range or significantly changed, the investigator deems it necessary to repeat the measurement, vital signs and 12-Lead ECG may be repeated twice, clinical laboratory tests [hematology, urinalysis, biochemistry and coagulation function test] may be repeated once):

    * Systolic blood pressure (SBP) ≥ 140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg after 5 minutes of supine rest;
    * Supine resting bradycardia (pulse heart rate [HR] <40 bpm) or a supine resting tachycardia (HR >100 bpm);
    * A corrected QT (QTc) interval of > 450 ms for males and > 470 ms for females (Fridericia's method);
    * Liver function: aspartate aminotransferase [AST], alanine transaminase [ALT], alkaline phosphatase [ALP], γ-glutamyl transferase [γ- GGT]) or total bilirubin (TBIL) >1.5 × upper limit of normal (ULN);
    * Renal function: creatinine clearance rate ≤80 mL/min (calculated based on Cockcroft-Gault formula);
    * Other laboratory parameters demonstrating clinically significant abnormalities, as determined by the investigator;
13. Known active infections, e.g., bacterial, fungal and viral infections, including:

    * Human immunodeficiency virus (HIV) infection: defined as HIV antibody positive;
    * Syphilis infection: defined as treponema pallidum antibody (TP-Ab) positive;
    * Active hepatitis B virus (HBV): defined as hepatitis B surface antigen (HBsAg) positive, Hepatitis B core antibody (HBcAb) positive and hepatitis B virus (HBV)-deoxyribonucleic acid (DNA) ≥ lab-specific ULN (for those with positive result on HBcAb or HBsAg, HBV DNA test will be performed and those with positive HBV DNA results will be excluded);
    * Active hepatitis C virus (HCV): defined as HCV antibody (HCV-Ab) positive and HCV-ribonucleic acid (RNA) positive, if HCV-Ab positive and HCV RNA negative can be considered as eligible at the discretion of the Investigator;
14. Has donated blood or plasma within 30 days prior to screening or had a loss of whole blood of more than 500 mL within the 30 days prior to screening, or receipt of a blood transfusion within one year prior to screening;
15. The subject has difficulty in swallowing oral medications;
16. Inability to be venipunctured and/or tolerate venous access; Any conditions which would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of VG290131 by TEAEs | From admission to discharge, up to 12 days.
  To evaluate the safety and tolerability of VG290131 after SAD and MAD doses to healthy volunteers by assessing the incidence, severity, and causality of treatment-emergent adverse events (TEAEs).
To evaluate the safety and tolerability of VG290131 by 12-Lead ECG | From admission to discharge, up to 12 days.
  To evaluate the safety and tolerability of VG290131 after SAD and MAD doses to healthy volunteers by assessing the number and percentage of subjects with clinically significant changes in 12-Lead ECG (RR, PR, QRSD, QT, and QTc).
To evaluate the safety and tolerability of VG290131 by vital signs | From admission to discharge, up to 12 days.
  To evaluate the safety and tolerability of VG290131 after SAD and MAD doses to healthy volunteers by assessing the number and percentage of subjects with clinically significant changes in vital signs (Blood pressure, heart rate, body temperature, and respiration rate).
To evaluate the safety and tolerability of VG290131 by physical examinations | From admission to discharge, up to 12 days.
  To evaluate the safety and tolerability of VG290131 after SAD and MAD doses to healthy volunteers by assessing the number and percentage of subjects with clinically significant changes in physical examinations (Skin and mucosa, lymph nodes, head, eyes, ears, nose, and throat (HEENT), chest, abdomen, spine and limbs, musculoskeletal system, and nervous system).
To evaluate the safety and tolerability of VG290131 by clinical laboratory tests | From admission to discharge, up to 12 days.
  To evaluate the safety and tolerability of VG290131 after SAD and MAD doses to healthy volunteers by assessing the number and percentage of subjects with clinically significant changes in clinical laboratory tests (hematology, coagulation, biochemistry and urine analysis).

SECONDARY OUTCOMES:
To evaluate PK parameter Cmax of VG290131 after a single dose | From admission to discharge, up to 12 days.
  Cmax of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter Tmax of VG290131 after a single dose | From admission to discharge, up to 12 days.
  Tmax of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter AUC0-t of VG290131 after a single dose | From admission to discharge, up to 12 days.
  AUC0-t of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter AUC0-inf of VG290131 after a single dose | From admission to discharge, up to 12 days.
  AUC0-inf of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter t1/2 of VG290131 after a single dose | From admission to discharge, up to 12 days.
  t1/2 of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter CL/F of VG290131 after a single dose | From admission to discharge, up to 12 days.
  CL/F of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter Vz/F of VG290131 after a single dose | From admission to discharge, up to 12 days.
  Vz/F of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter MRT of VG290131 after a single dose | From admission to discharge, up to 12 days.
  MRT of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter λz of VG290131 after a single dose | From admission to discharge, up to 12 days.
  λz of VG290131 under fasted and fed conditions will be calculated after a single dose.
To evaluate PK parameter Cmax,ss of VG290131 after multiple doses | From admission to discharge, up to 12 days.
  The maximum observed concentration at steady state (Cmax,ss) of VG290131 will be calculated after multiple doses from Day 1 to Day 7.
To evaluate PK parameter Cmin,ss of VG290131 after multiple doses | From admission to discharge, up to 12 days.
  The minimum observed concentration at steady state (Cmin,ss) of VG290131 will be calculated after multiple doses from Day 1 to Day 7.
To evaluate PK parameter Cav,ss of VG290131 after multiple doses | From admission to discharge, up to 12 days.
  The average concentration during a dosing interval at steady state (Cav,ss) of VG290131 will be calculated after multiple doses from Day 1 to Day 7.
To evaluate PK parameter AUCss of VG290131 after multiple doses | From admission to discharge, up to 12 days.
  The area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) of VG290131 will be calculated after multiple doses from Day 1 to Day 7.
To evaluate PK parameter Rac of VG290131 after multiple doses | From admission to discharge, up to 12 days.
  The accumulation ratio (Rac) of VG290131 will be calculated after multiple doses from Day 1 to Day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia